CLINICAL TRIAL: NCT05664360
Title: Incidence and Outcomes of Emergency Department Patients Requiring Emergency General Surgery
Status: Completed | Type: Observational
Sponsor: University Hospital, Geneva (Other)
Responsible Party: Principal Investigator, Christophe Fehlmann, Principal Investigator, University Hospital, Geneva
Other Study IDs: EGS1
Record Dates: First submitted 2022-12-09; First posted 2022-12-23 (Actual); Last update posted 2022-12-23 (Actual); Status verified 2022-12

CONDITIONS: Emergency General Surgery
MeSH Terms: interventions — Aging

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- ED patients
  Interventions: Other: Age (young versus older)

INTERVENTIONS:
Other: Age (young versus older) — Age

SUMMARY:
The objectives of this study were (1) to estimate the incidence of emergency general surgery in a Swiss University Hospital, (2) to describe the characteristics and outcomes of patients undergoing such interventions, and (3) to study the impact of age on the outcomes.

ELIGIBILITY:
Inclusion Criteria:

- consecutive patients visiting the emergency department

Exclusion Criteria:

* admitted primarily for a psychiatric reason
* left without consultation

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients visiting the emergency department
Sampling Method: Probability Sample
Enrollment: 310914 (Actual)
Dates: Start 2015-01-01 (Actual); Primary Completion 2022-03-15 (Actual); Study Completion 2022-03-15 (Actual)

PRIMARY OUTCOMES:
Incidence of emergency general surgery | Day 3
  Emergency general surgery following ED visit

SECONDARY OUTCOMES:
Admission to intensive care unit rate | During index hospitalization
  Admission to intensive care unit
ICU length of stay | During index hospitalization
  Number of days spent in the ICU during hospital stay
30-day mortality rate | 30 days
  30-day mortality
90-day mortality rate | 90 days
  90-day mortality
One-year mortality rate | One year
  One-year mortality
Hospital length of stay | During index hospitalization
  Hospital length of stay
Rate of patient dependent at discharge | Hospital discharge
  Dependent at discharge

CONTACTS AND LOCATIONS:
Overall Officials: Christophe A Fehlmann, MD, Principal Investigator — Genava University Hospitals

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Analytic Code
Time Frame: As soon as published
Access Criteria: Without restriction
URL: https://www.doi.org/10.17605/OSF.IO/TRU4N

REFERENCES:
- Available data/document: Individual Participant Data Set — https://www.doi.org/10.17605/OSF.IO/TRU4N